CLINICAL TRIAL: NCT04766021
Title: Mirabegron and Physiological Function in Cold Environments - Aim 1
Brief Title: Mirabegron and Physiological Function in Cold Environments
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Office of Naval Research (ONR) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Blair D. Johnson, PhD, Associate Professor School of Public Health, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2011690870; Aim 1
Record Dates: First submitted 2021-02-09; First posted 2021-02-23 (Actual); Results first posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Resting Energy Expenditure; Thermogenesis; Brown Adipose Tissue
MeSH Terms: interventions — mirabegron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Given once, followed by observation for 6 hours in a 20 degree Celsius (68 degree Fahrenheit) room
  Interventions: Drug: Placebo
- 100 mg Mirabegron (Experimental): Given once, followed by observation for 6 hours in a 20 degree Celsius (68 degree Fahrenheit) room
  Interventions: Drug: Mirabegron
- 150 mg Mirabegron (Experimental): Given once, followed by observation for 6 hours in a 20 degree Celsius (68 degree Fahrenheit) room
  Interventions: Drug: Mirabegron
- 200 mg Mirabegron (Experimental): Given once, followed by observation for 6 hours in a 20 degree Celsius (68 degree Fahrenheit) room
  Interventions: Drug: Mirabegron

INTERVENTIONS:
Drug: Mirabegron — Dose-response effect on thermogenesis
  Other Names: Myrbetriq
  Arms: 100 mg Mirabegron; 150 mg Mirabegron; 200 mg Mirabegron
Drug: Placebo — Placebo control condition
  Arms: Placebo

SUMMARY:
Many Navy diving operations are performed in cold water. Despite technical advances to improve thermal protection for cold water diving, these applications are cumbersome and do not provide complete thermal protection as thermal discomfort is subjectively reported by many Navy divers. Brown adipose tissue is highly thermogenic in humans. Therefore, activation of brown adipose tissue might improve cold water tolerance and lower thermal discomfort during cold water diving operations. Mirabegron is a beta-3-adrenergic receptor agonist that is used to treat overactive bladder. Beta-3-adrenergic receptors are located on the urinary bladder, gallbladder and brown adipose tissue. Recent evidence has demonstrated that acute mirabegron administration increases thermogenesis for ~3 hours in humans. However, it is currently not known which dose of mirabegron can increase thermogenesis for longer durations. It is also not known if mirabegron administration can improve cold water tolerance and thermal discomfort during cold water immersion. Finally, it is not known if mirabegron can increase thermogenesis during sympathetic stimulation. This project will fill these knowledge gaps by determining which dose of mirabegron administration will increase thermogenesis during 6 hours of a mild cold stress challenge. This study is part of a collection of studies that will show if mirabegron is a potential ergogenic aid that can be used to improve cold water tolerance in Navy divers which will ultimately improve the likelihood of successful missions.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, cross-over experimental design. Participants will be asked to complete 5 visits to the laboratory; one informed consent/screening visit and 4 study visits. On study visit days, participants will report to the laboratory following a 12-hour fast, and 24-hour abstention from exercise, caffeine, and alcohol. During the study visits, participants will be instrumented for skin temperature (12-sites: calf, shin, front of the thigh, back of the thigh, chest, upper back, forehead, lower back, abdomen, forearm, hand, and foot; iButtons) core temperature (rectal thermistor), indices of shivering (surface mechanomyography using triaxial accelerometers at 3 anatomic sites (chest, upper back, and thigh) and the bedside shivering assessment scale), brachial artery blood pressure (brachial artery auscultation), and heart rate (3-lead ECG). Thermal perceptions will be assessed using Likert scales for thermal discomfort and thermal sensation. Participants will be shirtless (sports bra for women) and will wear shorts throughout the study. After 20 minutes of quiet resting in the supine position, 5 minutes of baseline measurements will be taken, thermal perceptions and an infrared thermography image of the supraclavicular fossa will be obtained as an indicator of brown adipose tissue activation (6), and a whole blood sample will be obtained.

Participants will then ingest mirabegron (100 mg, 150 mg, or 200 mg) or placebo. Thirty minutes after mirabegron or placebo has been ingested, participants will enter the whole-body indirect calorimeter; the internal temperature of the calorimeter will be set to 20 degrees C (68 degrees F). This will elicit a mild cold stress over the 6 hours of observation in the whole-body indirect calorimeter. The whole-body indirect calorimeter provides an accurate and continuous measure of thermogenesis (in the form of energy expenditure) that can be used over long periods of time in a stable environment. The whole-body calorimeter is designed to perform human studies that are up to 48 hours in duration and contains a private washroom. While in the whole-body indirect calorimeter, participants will be instructed to be sedentary and will be allowed to watch television or read. In order to stay consistent between study visits, participants will be instructed to spend the same amount of time watching television or reading for each study visit. Every 30 minutes, we will record skin temperatures, core temperature, blood pressure, and heart rate. Thermogenesis will be determined by having participants lie supine for 30 minutes and resting energy expenditure will be calculated using the abbreviated Weir formula every hour (5). Thermal perceptions and an infrared thermography image will also be obtained at these time points. At approximately the midpoint of the 6-hour measurement period, participants will have the opportunity to use the restroom and an additional urine sample will be collected at this time. At the end of the 6-hour measurement period, participants will exit the whole-body indirect calorimeter and final measurements of skin temperature, core temperature, heart rate, and blood pressure will be obtained as well as a final infrared thermography image and a whole blood sample. After the experiment is complete, participants will be given a mylar blanket to re-warm themselves prior to leaving the laboratory.

Participants will be asked to return to the laboratory after 10-14 days to repeat the experiment until all 4 dosing conditions (placebo, 100 mg, 150 mg, and 200 mg of mirabegron) have been tested. Each participant's order of assignment to placebo or drug dosing over the 4 study visits will be randomly assigned.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* 18-40 years old
* Participate in 150 minutes or more of at least moderate intensity exercise per week during the previous 2 years

Exclusion Criteria:

* diagnosed autonomic disease
* diagnosed cardiovascular disease
* diagnosed metabolic disease
* diagnosed neurologic disease
* diagnosed endocrine disease
* diagnosed respiratory disease
* diagnosed liver dysfunction
* diagnosed kidney dysfunction
* Women who are pregnant or breastfeeding
* Individuals currently taking a medication (with the exception of birth control, including hormonal contraception) that cannot be safely discontinued for 5 biological half-lifes prior to each study visit based on consultation with the study physician.
* Current tobacco or electronic cigarette use or consistent use within the last 1 year

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Blair D Johnson, PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a repeated measures study design. 30 subjects provided written informed consent. Of these subjects: 9 voluntarily withdrew (4 provided no reason, 5 withdrew due to time commitment); 10 met exclusion criteria; 11 completed the informed consent/screening visit. All 11 subjects that completed the informed consent/screening visit also completed all four arms of the study.
Groups:
- Randomized: Placebo, 100 mg Mirabegron, 150 mg Mirabegron, 200 mg Mirabegron: Study drug/placebo given at baseline, followed by observation for 6 hours in a 20 degree Celsius (68 degree Fahrenheit) room
  Placebo: Four encapsulated placebo tablets 100 mg mirabegron: Two 50 mg mirabegron encapsulated tablets and two placebo encapsulated tablets 150 mg mirabegron: Three 50 mg mirabegron encapsulated tablets and one placebo encapsulated tablet 200 mg mirabegron: Four 50 mg mirabegron encapsulated tablets and one placebo encapsulated tablet
Period: Informed Consent/Screening Visit
Arm/Group | Randomized: Placebo, 100 mg Mirabegron, 150 mg Mirabegron, 200 mg Mirabegron
Started | 30
Completed | 11
Not Completed | 19
Not completed — Withdrawal by Subject | 9
Not completed — Met exclusion criteria | 10
Period: Interventions
Arm/Group | Randomized: Placebo, 100 mg Mirabegron, 150 mg Mirabegron, 200 mg Mirabegron
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Randomized: Placebo, 100 mg Mirabegron, 150 mg Mirabegron, 200 mg Mirabegron: Placebo: given once Mirabegron: 100 mg given once Mirabegron: 150 mg given once Mirabegron: 200 mg given once
  Participants completed each condition in a randomized order separated by 10-14 days. After placebo or mirabegron ingestion, participants were observed for 6 hours in a 20 degree Celsius (68 degree Fahrenheit) room.
Arm/Group | Randomized: Placebo, 100 mg Mirabegron, 150 mg Mirabegron, 200 mg Mirabegron
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 22 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 11
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 25 (4)

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Resting Energy Expenditure
Description: The cumulative resting energy expenditure will be calculated to reflect the cumulative effect of mirabegron over time.
Time Frame: 360 minutes
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | Placebo | 100 mg Mirabegron | 150 mg Mirabegron | 200 mg Mirabegron
Number analyzed (Participants) | 11 | 11 | 11 | 11
kcal | 456.4 (67.8) | 494.7 (75.7) | 481.3 (67.2) | 492.8 (69.8)

2. Secondary Outcome: Core Body Temperature
Description: Core Body temperature will be measured via rectal temperature during the experiment. The mean value was calculated.
Time Frame: Baseline and every 30 minutes through 360 minutes
Measure: Mean (Standard Deviation); unit: degrees C
Arm/Group | Placebo | 100 mg Mirabegron | 150 mg Mirabegron | 200 mg Mirabegron
Number analyzed (Participants) | 11 | 11 | 11 | 11
degrees C | 36.87 (0.03) | 36.78 (0.02) | 36.85 (0.04) | 36.76 (0.06)

3. Secondary Outcome: Brown Adipose Tissue Activation
Description: Infrared thermography will be used to measure supraclavicular skin temperature as an estimate of brown adipose tissue activation. The mean value was calculated.
Time Frame: Baseline and hourly through 360 minutes
Measure: Mean (Standard Deviation); unit: degrees C
Arm/Group | Placebo | 100 mg Mirabegron | 150 mg Mirabegron | 200 mg Mirabegron
Number analyzed (Participants) | 11 | 11 | 11 | 11
degrees C | 34.56 (0.25) | 34.49 (0.23) | 34.45 (0.25) | 34.45 (0.27)

4. Secondary Outcome: Weighted Mean Skin Temperature
Description: Fourteen iButtons will be adhered to the skin using adhesive tape on the calf, shin, front thigh, back thigh, foot, chest, upper back, lower back, forearm, hand, forehead, fingertip, toetip, and abdomen area to measure weighted skin temperature. Temperature readings will be taken every 30 minutes during the experiment. The mean value was calculated.
Time Frame: Baseline and every 30 minutes through 360 minutes
Measure: Mean (Standard Deviation); unit: degrees C
Arm/Group | Placebo | 100 mg Mirabegron | 150 mg Mirabegron | 200 mg Mirabegron
Number analyzed (Participants) | 11 | 11 | 11 | 11
degrees C | 30.58 (0.29) | 30.64 (0.28) | 30.43 (0.35) | 30.75 (0.31)

5. Secondary Outcome: Heart Rate
Description: Heart rate will be obtained using a 3-lead electrocardiogram. The mean value was calculated.
Time Frame: Baseline and every 30 minutes through 360 minutes
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Placebo | 100 mg Mirabegron | 150 mg Mirabegron | 200 mg Mirabegron
Number analyzed (Participants) | 11 | 11 | 11 | 11
beats/minute | 64 (2) | 69 (3) | 67 (2) | 68 (4)

6. Secondary Outcome: Mean Arterial Pressure
Description: Blood pressure will be monitored using a cuff placed on the upper arm that is inflated and deflated periodically. The mean value was calculated.
Time Frame: Baseline and every 30 minutes through 360 minutes
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | 100 mg Mirabegron | 150 mg Mirabegron | 200 mg Mirabegron
Number analyzed (Participants) | 11 | 11 | 11 | 11
mmHg | 92.5 (1.8) | 94.4 (2.3) | 95.4 (2.6) | 95.0 (3.2)

7. Secondary Outcome: Relative Oxygen Consumption
Description: A pneumotach connected to a mouthpiece or facemask will be used to measure the flow of inspired and expired air. Expired gases will be sampled using oxygen and carbon dioxide sensors to determine oxygen consumption and carbon dioxide production. The mean value was calculated.
Time Frame: Baseline and every 30 minutes through 360 minutes
Measure: Mean (Standard Deviation); unit: ml O2 / kg body mass / minute
Arm/Group | Placebo | 100 mg Mirabegron | 150 mg Mirabegron | 200 mg Mirabegron
Number analyzed (Participants) | 11 | 11 | 11 | 11
ml O2 / kg body mass / minute | 3.59 (0.12) | 3.89 (0.20) | 3.83 (0.22) | 3.89 (0.18)

8. Secondary Outcome: Bedside Shivering Scale
Description: Two investigators will subjectively assess shivering by the participants using a Likert scale (range 0-3; 0 = none, 3 = Severe) and the scores will be averaged. The mean value was calculated.
Time Frame: Baseline and every 30 minutes through 360 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 100 mg Mirabegron | 150 mg Mirabegron | 200 mg Mirabegron
Number analyzed (Participants) | 11 | 11 | 11 | 11
units on a scale | 0.06 (0.22) | 0.04 (0.18) | 0.02 (0.11) | 0.03 (0.14)

9. Secondary Outcome: Thermal Comfort Scale
Description: Participants will complete a Likert scale to assess their thermal comfort (range: 1-4; 1 = comfortable, 4 = very uncomfortable).The mean value was calculated.
Time Frame: Baseline and every 30 minutes through 360 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 100 mg Mirabegron | 150 mg Mirabegron | 200 mg Mirabegron
Number analyzed (Participants) | 11 | 11 | 11 | 11
units on a scale | 2.1 (0.3) | 1.9 (0.3) | 1.9 (0.2) | 1.8 (0.2)

10. Secondary Outcome: Thermal Sensation Scale
Description: Participants will complete a Likert scale to assess their thermal sensation (range: 1-7; 1 = cold, 4 = neutral, 7 = hot). The mean value was calculated.
Time Frame: Baseline and every 30 minutes through 360 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 100 mg Mirabegron | 150 mg Mirabegron | 200 mg Mirabegron
Number analyzed (Participants) | 11 | 11 | 11 | 11
units on a scale | 2.4 (0.4) | 2.8 (0.3) | 2.7 (0.3) | 2.8 (0.3)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for each subject after informed consent was obtained and up to their study completion (up to 7 months).
Arm/Group | Placebo | 100 mg Mirabegron | 150 mg Mirabegron | 200 mg Mirabegron
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-29): https://cdn.clinicaltrials.gov/large-docs/21/NCT04766021/Prot_SAP_000.pdf
  • Informed Consent Form (2024-01-29): https://cdn.clinicaltrials.gov/large-docs/21/NCT04766021/ICF_001.pdf